CLINICAL TRIAL: NCT01641198
Title: Prospective Randomized Clinical Trial Comparing Quantitative Osseous Healing of Acid Etched and Machined Titanium Implant Fixtures After 12 and 24 Months, and at 15-20 Years of Function With Full Arch Fixed Mandibular Prostheses.
Brief Title: An Implant With an Acid-etched Fixture Surface and Internal-hex Collar May Achieve Greater Osseointegration.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: Medical Research Council of Canada, FRSQ, CoreVent, Université de Montréal (Unknown)
Responsible Party: Principal Investigator, Aldo Joseph Camarda, Associate Professor, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-069-CERES-D
Record Dates: First submitted 2012-07-06; First posted 2012-07-16 (Estimated); Results first posted 2019-01-16 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Jaw, Edentulous; Dental Implant
Keywords: Dental Implants Microtextured Fixture Machined Collar Bone
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Configuration 1 (Active Comparator): Device placement: B (Brånemark) at two sites, SW (Swede-Vent) at two sites, SC (Screw-Vent) at one site
  Interventions: Device: Configuration 1
- Configuration 2 (Experimental): Device placement: B (Brånemark) at one site, SW (Swede-Vent) at two sites, SC (Screw-Vent) at two sites
  Interventions: Device: Configuration 2
- Configuration 3 (Experimental): Device placement: B (Brånemark) at two sites, SW (Swede-Vent) at one site, SC (Screw-Vent) at two sites
  Interventions: Device: Configuration 3

INTERVENTIONS:
Device: Configuration 1 — B placed at sites 2 and 5, SW placed at sites 1 and 4, SC placed at site 3
  Arms: Configuration 1
Device: Configuration 2 — B placed at site 3, SW placed at sites 2 and 5, SC placed at sites 1 and 4
  Arms: Configuration 2
Device: Configuration 3 — B placed at sites 1 and 4, SW placed at site 3, SC placed at sites 2 and 5
  Arms: Configuration 3

SUMMARY:
Brånemark System® dental implant osseointegration was introduced clinically in 1965 as a novel approach to the replacement of missing teeth. Although this implant's traditional machined screw-shaped surface had excellent, well-documented short- and long-term osseointegration success, newer implant designs were introduced that could enhance biological fusion of the implant to jaw bones, allowing more rapid restoration and function. It was also claimed that such implants could lead to less bone loss with function. One such implant, Screw-Vent®, had a macrostructure very similar to that of the Brånemark implant, except that it's fixture surface was acid-etched which could enhance biological osseointegration. It also had a longer narrower smooth internal-hex interlocking flat collar that could better resist occlusal forces, leading to even less bone loss according to the manufacturer. However, no well-controlled clinical studies existed in 1990 that supported these claims. This study was undertaken, therefore, to first compare the Brånemark implant with another implant, Swede-Vent®, a copy of the Brånemark implant except for its fixture surface that was identically acid-etched as that of Screw-Vent by the same manufacturer. The effect on bone healing could then be compared between Brånemark's machined and Swede-Vent's acid-etched surfaces in the short- and long-terms. Our hypothesis was that the microtextured Swede-Vent fixture would lead to greater bone preservation. Since Screw-Vent's fixture surface was identically acid-etched as that of Swede-Vent by the same manufacturer, we could then evaluate the effect on bone healing of Screw-Vent's collar and the shorter wider machined smooth external-hex flat collar of Swede-Vent (identical to that of Brånemark). All three 2-part platform-matched parallel-wall implants were made of commercially pure titanium, had a very similar fixture macro-design, were approved by the Food and Drug Administration (USA) and Health and Welfare Canada, and were commercially available in North America. Brånemark is still available, but with an oxidized microtextured fixture surface and a shortened machined smooth external-hex flat collar. Screw-Vent is still available with its microtextured fixture surface, but its machined smooth internal-hex flat collar has also been substantially shortened. Swede-Vent is no longer available.

DETAILED DESCRIPTION:
This prospective randomized long-term superiority clinical trial tests the hypothesis that an implant with an acid-etched fixture surface and internal-hex machined flat collar results in greater bone preservation.

Age-eligible participants were recruited into this study between 1990 and 1992 from the external clinics of a university dental faculty and hospital affiliated dental department. Study was peer reviewed, had satisfied ethics committee's criteria for human clinical research, and was to take place at the university dental faculty and hospital affiliated department. Sixty participants were enrolled. The study's coordinator evaluated clinical charts to confirm that participants had satisfied the pre-determined inclusion criteria, and that registry operations, data collection, documentation and analysis followed established protocol.

A statistician who was not part of the research team prepared a sampling design that included three Configurations. Each Configuration contained five implants of the three types, thereby allowing an equal number of each implant type to be placed in a cyclical side-by-side rotating fashion at each of five sites between the mental foramen. Consequently, 100 implants of each of the three types were to be placed for a total of 300. However, two participants opted out before start of study so that 58 (30 women) received 290 implants, and each participant acted as their own control. A different identification number was placed on each participant's chart, and allocation concealment then allowed 20 participants to receive Configuration 1, 19 Configuration 2, and 19 Configuration 3. Configuration diagram (but not number) identifying the implant type and length to be placed at each site was stored inside each chart, and only shown to the operating team at surgery. Following restoration with a fixed complete dental prosthesis on the implants, each participant was examined and standardized peri-apical radiographs were taken of each implant after 12 and 24 months and at 15-20 years of function. Distance between first bone-to-implant contact point (fBIC) and crestal abutment-implant interface/microgap (MG) was measured at right and left sides of each abutment-implant surface on the radiographs by examiners who were not part of the research team. Mean fBIC-MG values were then calculated, documented and compared between Brånemark, Swede-Vent and Screw-vent at the three intervals.

Assessment was based on intention to treat. Inter and intra-examiner reliability of measurements was assessed using Intraclass Correlation Coefficient and Bland-Altman Repeatability. Statistical analysis was based on the mixed linear model that included fixed effects of time, implant position, implant configuration, implant type (and implant length as a covariate effect). Position and time were repeated within participants, and Shapiro-Wilk Test was applied to verify that data was following normal distribution. Bonferroni correction was used for pairwise comparisons, and a p value of <0.05 was considered significant. Confidence Interval was established at 2-sided 95% Confidence Level. All statistical analyses were performed using Statistical Package for the Social Sciences (SPSS) Version 23® (IBM Corp, Armonk US).

The following were consulted in order to utilize standardized descriptive terms.

American Society of Anesthesiologists Physical Status Classification System (1963) was used to classify each participant's physical health as Class 1 (obligatory).

Lekholm-Zarb Classification System (1987) was used to classify each participant's quality (density) of mandibular bone as Types 2 and 3 (obligatory).

Salzman Skeletal Bone Intermaxillary Classification System (1966) was used to classify each participant's profile skeletal relationship between maxilla and mandible as Class 1 (obligatory).

American Psychological Association (APA) Publication Manual (2001, fifth edition, Washington, DC) was used to describe certain participant baseline demographic characteristics.

ELIGIBILITY:
No systemic disease (ASA Class 1)

Aged between 25 and 56 years

Non-smoking

No Temporomandibular Joint (TMJ) disorder or other facial pain

Wearing of complete maxillary and mandibular removable prostheses for at least one year

Skeletal Class 1 inter-maxillary relationship

Type 2 and/or Type 3 mandibular bone quality

Possess at least 1 cm of bone height between the superior and inferior cortical tables and at least 6 mm of bucco-lingual bone width between mental foramen

Specifically requesting a fixed full arch dental prosthesis over the implants and a conventional full arch removable maxillary prosthesis

Accepting to sign informed consent documents.

Ages: 25 Years to 56 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 1992-03 (Actual); Primary Completion 1998-03-24 (Actual); Study Completion 2013-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Milot, DMD,MSD, Principal Investigator — Université de Montréal; Hugo Ciaburro, DMD, MSc, Principal Investigator — Université de Montréal; Aldo-Joseph Camarda, DDS, MSc, Principal Investigator — Université de Montréal
Locations (1):
- Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 1990 - 1992
Pre-assignment Details: Sixty participants were recruited; however, two participants opted out prior to informed consent and random assignment to an arm.
Units Other Than Participants: Implants
Groups:
- Configuration 1: Surgical placement of devices (implants): B at sites 2 and 5, SW at sites 1 and 4, SC at site 3
- Configuration 2: Surgical placement of devices (implants): B at site 3, SW at sites 2 and 5, SC at sites 1 and 4
- Configuration 3: Surgical placement of devices (implants): B at sites 1 and 4, SW at site 3, SC at sites 2 and 5
Period: After 12 Months of Function
Arm/Group | Configuration 1 | Configuration 2 | Configuration 3
Started | 20; 100 Implants | 19; 95 Implants | 19; 95 Implants
Completed | 16; 67 Implants (Participants: 3 interval violation, 1 protocol violation. Implants: 13 bone loss not measurable) | 16; 77 Implants (Participants: 2 interval violation, 1 adverse event. Implants: 3 bone loss not measurable) | 17; 82 Implants (Participants: 2 interval violation. Implants: 3 bone loss not measurable)
Not Completed | 4; 33 Implants | 3; 18 Implants | 2; 13 Implants
Not completed — Lost to Follow-up | 3 | 2 | 2
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0
Period: After 24 Months of Function
Arm/Group | Configuration 1 | Configuration 2 | Configuration 3
Started | 16; 67 Implants | 16; 77 Implants | 17; 82 Implants
Completed | 12; 57 Implants (Participants: 4 interval violation. Implants: 3 bone loss not measurable) | 7; 35 Implants (Participants: 9 interval violation) | 11; 53 Implants (Participants: 6 interval violation. Implants: 2 bone loss not measurable)
Not Completed | 4; 10 Implants | 9; 42 Implants | 6; 29 Implants
Not completed — Lost to Follow-up | 4 | 9 | 6
Period: At 15-20 Years of Function
Arm/Group | Configuration 1 | Configuration 2 | Configuration 3
Started | 12; 57 Implants | 7; 35 Implants | 11; 53 Implants
Completed | 6; 30 Implants (Participants: 5 interval violation, 1 death) | 6; 30 Implants (Participants: 1 interval violation) | 9; 45 Implants (Participants: 1 interval violation, 1 death)
Not Completed | 6; 27 Implants | 1; 5 Implants | 2; 8 Implants
Not completed — Lost to Follow-up | 5 | 1 | 1
Not completed — Death | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Units Other Than Participants: Implants
Groups:
- Total: Total of all reporting groups
Arm/Group | Configuration 1 | Configuration 2 | Configuration 3 | Total
Number analyzed (Participants) | 20 | 19 | 19 | 58
Number analyzed (Implants) | 100 | 95 | 95 | 290
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (5.3) | 45.5 (5.6) | 44.8 (6.1) | 45.2 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 10 | 30
  Male | 10 | 9 | 9 | 28
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 20 | 19 | 19 | 58
Number of Participants with Health Status ASA Classification 1 [Count of Participants; unit: Participants] — Health status for all participants must be American Society of Anesthesiologists (ASA) Classification 1: participant has no systemic medical disease.
  Participants | 20 | 19 | 19 | 58
Number of Participants with Mandibular bone classification types 2 & 3 [Count of Participants; unit: Participants] — Mandibular bone density for all participants must be Lekholm-Zarb Classification Type 2 and 3: mandible must have a thick or thin layer of cortical bone that surrounds a core dense trabecular bone of favorable strength.
  Participants | 20 | 19 | 19 | 58
Removable complete dental prostheses obligatory [Count of Participants; unit: Participants] — All participants must have been wearing complete removable dentures for at least 1 year
  Participants | 20 | 19 | 19 | 58
Specifically requesting a complete lower prosthesis on implants [Count of Participants; unit: Participants] — All participants must have requested a complete fixed denture over the implants and a complete removable upper denture
  Participants | 20 | 19 | 19 | 58
Accepting to sign informed consent documents [Count of Participants; unit: Participants] — All participants must accept to sign informed consent documentation
  Participants | 20 | 19 | 19 | 58

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Quantitative Bone Healing
Description: Distance between first bone-to-implant contact point (fBIC) and microgap (MG) placed at the crest was measured at the right and left sides of each implant-abutment complex on periapical radiographs taken of each implant. Measurements were taken and recorded after 12 months of function. Mean fBIC-MG values were calculated, recorded and compared between B and SW, between B and SC and between SW and SC for Configuration 1, Configuration 2 and Configuration 3
Time Frame: After 12 months of function
Population: Reasons for decrease in population number: 7 did non-respect interval follow up protocol, 1 adverse event, 1 protocol violation. Reasons for decrease in number of units (implants): radiographs did not allow precise location of first bone-to-implant contact point (fBIC) and microgap (MG) due to technical reasons for 19 implants
Measure: Mean (Standard Error); unit: mm
Units Other Than Participants: Implants.
Arm/Group | Configuration 1 | Configuration 2 | Configuration 3
Number analyzed (Participants) | 16 | 16 | 17
Number analyzed (Implants.) | 67 | 77 | 82
mm | -1.18 (0.15) | -1.01 (0.16) | -0.91 (0.17)
Statistical Analysis 1: Comparison: Configuration 1 vs Configuration 2 vs Configuration 3; Mean bone change between B and SW estimated with the mixed linear model (mean±SE, 95% CI); Test type: Superiority; p < 0.05, Mixed Models Analysis — Statistical analysis was based on the mixed linear model with the level of significance set at p<0.05 and Bonferroni correction for pairwise comparisons; Mixed linear model with effects of time, implant position, implant configuration, implant type (and implant length as a covariate effect); Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.59 to 0.01], Standard Error of Mean 0.115
Statistical Analysis 2: Comparison: Configuration 1 vs Configuration 2 vs Configuration 3; Mean bone change between B and SC estimated with the mixed linear model (mean±SE, 95% CI); Test type: Superiority; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.39, 95% CI 2-sided [0.09 to 0.69], Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: Configuration 1 vs Configuration 2 vs Configuration 3; Mean bone change between SW and SC estimated with the mixed linear model (mean±SE, 95% CI); Test type: Superiority; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.685, 95% CI 2-sided [-0.98 to -0.39], Standard Error of Mean 0.115

2. Primary Outcome: Comparison of Quantitative Bone Healing
Description: Distance between first bone-to-implant contact point (fBIC) and microgap (MG) placed at the crest is measured at the right and left sides of each implant-abutment complex on periapical radiographs taken of each implant. Measurements were taken and recorded after 24 months of function. Mean fBIC-MG values were calculated, recorded and compared between B and SW, between B and SC and between SW and SC for Configuration 1, Configuration 2 and Configuration 3
Time Frame: After 24 months of function
Population: Reasons for decrease in the number of participants: 19 did not respect follow up interval. Reasons for decrease in number of units (implants): radiographs did not allow precise location of first bone-to-implant contact point (fBIC) and microgap (MG) due to technical reasons for 5 implants
Measure: Mean (Standard Error); unit: mm
Units Other Than Participants: implants
Arm/Group | Configuration 1 | Configuration 2 | Configuration 3
Number analyzed (Participants) | 12 | 7 | 11
Number analyzed (implants) | 57 | 35 | 53
mm | -1.16 (0.18) | -0.87 (0.23) | -1.33 (0.18)
Statistical Analysis 1: Comparison: Configuration 1 vs Configuration 2 vs Configuration 3; Mean bone change between B and SW estimated with the mixed linear model (mean±SE, 95% CI); Test type: Superiority; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.47 to 0.13], Standard Error of Mean 0.135
Statistical Analysis 2: Comparison: Configuration 1 vs Configuration 2 vs Configuration 3; Mean bone change between B and SC estimated with the mixed linear model (mean±SE, 95% CI); Test type: Superiority; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.56, 95% CI 2-sided [0.26 to 0.85], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: Configuration 1 vs Configuration 2 vs Configuration 3; Mean bone change between SW and SC estimated with the mixed linear model (mean±SE, 95% CI); Test type: Superiority; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.725, 95% CI 2-sided [-1.02 to -0.43], Standard Error of Mean 0.135

3. Primary Outcome: Comparison of Quantitative Bone Healing
Description: Distance between first bone-to-implant contact point (fBIC) and microgap (MG) placed at the crest is measured at the right and left sides of each implant-abutment complex on periapical radiographs taken of each implant. Measurements were taken and recorded at 15 to 20 years of function. Mean fBIC-MG values were calculated, recorded and compared between B and SW, between B and SC and between SW and SC for Configuration 1, Configuration 2 and Configuration 3
Time Frame: At 15-20 years of function
Population: Reasons for decrease in the number of participants: 7 did not respect follow up interval, 2 unrelated deaths
Measure: Mean (Standard Error); unit: mm
Units Other Than Participants: implants
Groups:
- Configuration 3: Surgical placement of devices (implants): B at sites1 and 4, SW at site 3, SC at sites 2 and 5
Arm/Group | Configuration 1 | Configuration 2 | Configuration 3
Number analyzed (Participants) | 6 | 6 | 9
Number analyzed (implants) | 30 | 30 | 45
mm | -1.32 (0.27) | -1.42 (0.33) | -1.54 (0.33)
Statistical Analysis 1: Comparison: Configuration 1 vs Configuration 2 vs Configuration 3; Mean bone change between B and SW estimated with the mixed linear model (mean±SE, 95% CI); Test type: Superiority; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-0.19 to 0.59], Standard Error of Mean 0.20
Statistical Analysis 2: Comparison: Configuration 1 vs Configuration 2 vs Configuration 3; Mean bone change between B and SC estimated with the mixed linear model (mean±SE, 95% CI); Test type: Superiority; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.83, 95% CI 2-sided [0.45 to 1.22], Standard Error of Mean 0.20
Statistical Analysis 3: Comparison: Configuration 1 vs Configuration 2 vs Configuration 3; Mean bone change between SW and SC estimated with the mixed linear model (mean±SE, 95% CI); Test type: Superiority; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.635, 95% CI 2-sided [-1.01 to -0.26], Standard Error of Mean 0.20

ADVERSE EVENTS:
Time Frame: Adverse data collection after 12 and 24 months, and 15-20 years of function
Arm/Group | Configuration 1 | Configuration 2 | Configuration 3
All-Cause Mortality (participants affected / at risk) | 1/20 | 0/19 | 1/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Configuration 1 (N=20) | Configuration 2 (N=19) | Configuration 3 (N=19)
Loss of jaw implant (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated jaw fracture with loss of one implant

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No